CLINICAL TRIAL: NCT02480010
Title: An Open Label, Phase II, Multicenter Study to Evaluate the Efficacy and Safety of a Recombinant Humanized Antibody to HER2 (Pertuzumab) Administered Every 3 Weeks to Patients With Hormone-Refractory Prostate Cancer Who Have Not Been Treated With Chemotherapy
Brief Title: A Study of Pertuzumab in Participants With Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated at the time of interim analysis since none of the participants showed a PSA response.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO17004
Record Dates: First submitted 2015-06-05; First posted 2015-06-24 (Estimated); Results first posted 2015-09-18 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pertuzumab

ARMS (2):
- Pertuzumab 1050 mg (Cohort B) (Experimental): Participants in Cohort B will receive 1050 mg pertuzumab via IV infusion on Day 1 of each 3-week cycle. At the end of 3 treatment cycles, response will be evaluated to determine whether additional participants will be enrolled for treatment. If a second stage of enrollment occurs, participants may continue treatment until disease progression or unacceptable toxicity.
  Interventions: Drug: Pertuzumab
- Pertuzumab 420 mg (Cohort A) (Experimental): Participants in Cohort A will receive an IV loading dose of 840 milligrams (mg) pertuzumab followed by 420 mg via IV infusion on Day 1 of each 3-week cycle. At the end of 3 treatment cycles, response will be evaluated to determine whether additional participants will be enrolled for treatment. If a second stage of enrollment occurs, participants may continue treatment until disease progression or unacceptable toxicity.
  Interventions: Drug: Pertuzumab

INTERVENTIONS:
Drug: Pertuzumab — Participants will receive pertuzumab on Day 1 of each 3-week cycle. In Cohort A, an 840-mg loading dose will be administered prior to the 420-mg IV infusion. In Cohort B, the 1050-mg IV infusion will be administered with no loading dose.
  Other Names: Perjeta

SUMMARY:
This study will evaluate the efficacy and safety of intravenous (IV) pertuzumab in participants with hormone-refractory prostate cancer who have had no previous chemotherapy. Participants will be enrolled in two stages, the first (Cohort A) at a lower 420-mg dose and the second (Cohort B) at a higher 1050-mg dose based upon observations in Cohort A. Up to 50 participants may enter either cohort, for a total enrollment between 46 and 73 participants across 9 study centers.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than (>) 18 years of age
* Histologically documented adenocarcinoma of the prostate resistant to hormone therapy, progressed at 4 to 6 weeks following anti-androgen withdrawal
* Prostate-specific antigen (PSA) values at least 20 ng/mL among those with asymptomatic or mildly symptomatic disease
* Karnofsky performance status (KPS) at least 80 percent (%)
* Castrate testosterone less than (<) 50 ng/dL
* Life expectancy at least 12 weeks
* Left ventricular ejection fraction (LVEF) at least 50%
* Adequate hematologic, hepatic, and renal function

Exclusion Criteria:

* Prior chemotherapy, radionucleotide therapy, or immunotherapy for prostate cancer
* Systemic corticosteroids within 1 month prior to Screening
* Bisphosphonates within 6 months, narcotic analgesics within 2 weeks, or any investigational agent with 28 days of study drug
* Prior cumulative doxorubicin dose of > 360 mg/m^2 or equivalent
* Central nervous system (CNS) or pulmonary metastases
* Other malignancies, except adequately treated basal or squamous cell skin cancer
* Significant cardiovascular disease
* Active/uncontrolled concurrent illness or infection
* Major surgery or traumatic injury within 4 weeks of study drug

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2003-09; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (11):
- France (2):
  - Lyon
  - Montpellier
- Berlin, Germany
- Italy (2):
  - Parma
  - Roma
- Rotterdam, Netherlands
- Spain (2):
  - Barcelona
  - Valencia
- United Kingdom (3):
  - Cardiff
  - Sutton
  - Weston-super-Mare

RESULTS

PARTICIPANT FLOW:
Groups:
- Pertuzumab 420 Milligrams (mg) - Cohort A: Participants in Cohort A received an intravenous (IV) loading dose of 840 mg pertuzumab on Day 1 of Cycle 1 (3-week cycles); from Cycle 2 onwards, participants received IV infusions of 420 mg on Day 1. Treatment continued for a maximum of 36 cycles or until study termination.
- Pertuzumab 1050 mg - Cohort B: Participants in Cohort B received 1050 mg pertuzumab as an IV infusion on Day 1 of each 3-week cycle for a maximum of 36 cycles or until study termination.
Period: Overall Study
Arm/Group | Pertuzumab 420 Milligrams (mg) - Cohort A | Pertuzumab 1050 mg - Cohort B
Started | 35 | 33
Completed | 0 | 0
Not Completed | 35 | 33
Not completed — Adverse Event | 3 | 1
Not completed — Death | 1 | 0
Not completed — Insufficient therapeutic response | 31 | 29
Not completed — Refused Treatment | 0 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population consisted of all participants enrolled and who received at least one dose of study medication.
Groups:
- Pertuzumab 420 mg - Cohort A: Participants in Cohort A received an IV loading dose of 840 mg pertuzumab on Day 1 of Cycle 1 (3-week cycles); from Cycle 2 onwards, participants received IV infusions of 420 mg on Day 1. Treatment continued for a maximum of 36 cycles or until study termination.
- Total: Total of all reporting groups
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B | Total
Number analyzed (Participants) | 35 | 33 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (7.45) | 71.2 (6.01) | 71.0 (6.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 35 | 33 | 68

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Confirmed, Objective Response, Non-Response or Progressive Disease by PSA Levels Within the First 24 Weeks of Treatment With Pertuzumab
Description: Objective PSA response rate was determined according to Prostate Specific Antigen Working Group (PSAWG) guidelines. All participants achieving a drop in PSA of greater than or equal to (≥) 50 percent (%) from baseline (confirmed with a second value at least 4 weeks later) fulfilled the criteria of a PSA response. The confirmatory second value had to be at least 50% lower than baseline, but could be higher than the first drop in PSA. Confirmatory value could not be 50% higher compared to first drop in PSA. The date of response was the date the first 50% (or greater) decline was observed. Progressive disease (PD) was defined by a minimum of three consecutive serum PSA measurements obtained at least 7 days apart within the previous 3 months of start of trial, which documented progressively increasing values. Non-response was defined as neither PD nor Response.
Time Frame: Screening, Every 3 weeks up to Week 24
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 35 | 33
percentage of participants
  Objective response | 0.0 | 0.0
  Non-response | 34.3 | 30.3
  PD | 65.7 | 66.7
  Missing | 0.0 | 3.0

2. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression was defined by time in weeks from start of therapy to the onset of the earliest of the following events. 1) PSA progression as defined by the PSAWG, 2) Evidence of disease progression according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria 3) One bone scan at least 6 months subsequent to baseline demonstrating 2 or more new skeletal lesions and 4) An event due to metastatic prostate cancer requiring intervention.
Time Frame: Screening, Every 3 weeks up to a maximum of 18 months
Population: ITT population
Measure: Median (Full Range); unit: weeks
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 34 | 30
weeks | 5.6 [2.8 to 20.9] | 6.1 [2.7 to 17.9]

3. Secondary Outcome: Percentage of Participants With Objective Response (Complete Response [CR] or Partial Response [PR]) by Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Overall objective response by RECIST criteria (CR or PR) was to be defined for participants who had measurable disease at baseline or developed new lesions post-baseline. The longest diameter only for all target lesions was measured and the following responses recorded: CR: disappearance of all target lesions. PR: at least a 30% decrease in the sum of the longest diameter as compared to the baseline sum longest diameter.
Time Frame: Screening, Weeks 6, 12, 24, 36 and 48
Population: This analysis was only planned if either cohort went to full recruitment. Analysis of this outcome in a small number of participants would have high variability and also unlikely to be relevant if safety and tolerability criteria were not met.
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Response
Description: Time to response was the date of the first documentation of PSA response.
Time Frame: Screening, Every 3 weeks for a maximum of 18 months
Population: as for outcome 3
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Duration of Response According to PSA Levels
Description: Duration of PSA Response was measured from first 50% decline in PSA compared to baseline until the time at which there was an increase of ≥50% from the PSA nadir, provided the absolute increase was at least 5 nanograms per milliliter (ng/ml). The increase must have been confirmed by a second consecutive measurement that was at least 50% above the nadir.
Time Frame: Baseline, Every 3 weeks for a maximum of 18 months
Population: as for outcome 3
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Duration of Response According to RECIST Criteria
Description: For participants with measurable disease, duration of response was defined as first documentation of tumor response, either a PR or CR, to first documentation of PD or death. Participants who never progressed or died were censored at their last tumor measurement.
Time Frame: Baseline, Weeks 6, 12, 24, 36 and 48
Population: as for outcome 3
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants Without Progression
Description: Disease progression was defined as the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Non-progression included participants who had responded plus those who had not responded and not progressed within the first 3 cycles.
Time Frame: Screening, Weeks 3, 6, 9 and 12
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 35 | 33
percentage of participants | 20.0 | 18.2

8. Secondary Outcome: Time to Prostate Cancer Pain Progression
Description: Time to disease progression was defined by time in weeks from start of therapy to the onset of the earliest of the following events: 1) Opioid therapy, 2) Radiation therapy, 3) Glucocorticoid therapy, 4) Radionuclide therapy or 5) Chemotherapy.
Time Frame: Every 3 weeks up to a maximum of 18 weeks
Population: as for outcome 3
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the interval of time in weeks between start of treatment and day of death. Participants who did not die while being followed were censored at the last time that they were known to be alive.
Time Frame: Screening, Every 3 weeks up to a maximum of 18 months
Population: Data were not analyzed due to early termination of the study.
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Time to Treatment Failure
Description: Time to Treatment Failure was time to the first documentation of progressive disease, day of death while on study (or 30 days after withdrawing from the trial) or day of early discontinuation due to toxicity (adverse events or abnormal laboratory value), refusal of treatment/refusing to cooperate/withdrawing consent, insufficient therapeutic response, or failure to return, whichever is earliest, after the start of treatment. Participants who did not experience any of the above events while on study were censored on the day of their last PSA or tumor measurement, whichever was later.
Time Frame: Every 3 weeks up to a maximum of 18 weeks
Population: ITT Population
Measure: Median (Full Range); unit: days
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 35 | 33
days | 6.1 [2.8 to 20.9] | 6.1 [2.7 to 17.9]

11. Secondary Outcome: Change From Baseline in Bone Alkaline Phosphatase
Description: Bone alkaline phosphatase (BAP) is the bone-specific isoform of alkaline phosphatase. Serum Bone alkaline phosphatase is used to measure osteoporosis and is measured as units per liter (u/L).
Time Frame: Screening, Weeks 6, 12, 24, 36 and 48
Population: Data were not analyzed to due to early termination of the study.
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change From Baseline in N-Telopeptide
Description: In bone physiology, the N-terminal telopeptide (or more formally, amino-terminal collagen crosslinks, and known by the acronym NTX) is a telopeptide that can be used as a biomarker to measure the rate of bone turnover. NTX can be measured in the urine (uNTX) or serum (serum NTX).
Time Frame: Screening, Weeks 6, 12, 24, 36 and 48
Population: Data were not analyzed to due to early termination of the study.
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Area Under the Concentration Curve Extrapolated to Infinity (AUC0-Inf) of Pertuzumab
Description: The area under the plot of plasma concentration of drug against time after drug administration is defined as the area under the curve (AUC). The AUC0-infinity is calculated from time 0 (prior to administration of medication) to infinity (the time of complete elimination of the drug). The AUC is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption. AUC is measured as micrograms times days per milliliter (µg*day/mL)
Time Frame: Cycles 1 and 2 (Weeks 3 and 6): predose (immediately prior to infusion) and within 15 minutes following the end of the infusion on Day 1, Day 8, and Day 15. Cycle 3 (Week 9) and beyond: predose and within 15 minutes following end of infusion on Day 1
Population: ITT Population; Only participants with non-missing data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*day/mL
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 35 | 31
µg*day/mL | 3488 (44) | 5097 (71)

14. Secondary Outcome: AUC to Last Measurable Concentration (AUC0-last) of Pertuzumab
Description: The AUC0-last is calculated from time 0 (prior to administration of medication) to last measured data point. The AUC is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption.
Time Frame: as for outcome 13
Population: ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg*day/mL
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 35 | 33
µg*day/mL | 2305 (22) | 2626 (28)

15. Secondary Outcome: Maximum Plasma Concentration of Pertuzumab
Description: Cmax is the maximum (or peak) plasma concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administered and prior to the administration of a second dose. Cmax is measured as micrograms per mL (μg/mL).
Time Frame: as for outcome 13
Population: ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 35 | 33
μg/mL | 255 (23) | 294 (24)

16. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Pertuzumab
Description: Cmax refers to the maximum (or peak) plasma concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administered and prior to the administration of a second dose. tmax is the time at which the Cmax is observed.
Time Frame: Cycles 1 and 2 (Weeks 3 and 6): predose (immediately prior to infusion) and within 15 minutes following the end of the infusion on Day 1 and on Days 8 and 15, Cycle 3 (Week 9) and beyond: predose and within 15 minutes following end of infusion on Day 1
Population: ITT Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 35 | 33
days | 0.073 (11) | 0.074 (6)

17. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of Pertuzumab
Description: t1/2 is the time in days required for the concentration of the drug to reach half of its original value
Time Frame: as for outcome 13
Population: ITT Population; Only participants with non-missing data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 35 | 31
days | 13.7 (39) | 19.3 (69)

18. Secondary Outcome: Serum Clearance of Pertuzumab
Description: Clearance (expressed as volume/time) describes the removal of drug from a volume of plasma in a given unit of time (drug loss from the body). It is measured as milliliters per day (mL/day).
Time Frame: as for outcome 13
Population: ITT Population; Only participants with non-missing data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/day
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 35 | 31
mL/day | 270 (29) | 253 (35)

19. Secondary Outcome: Volume of Distribution at Steady State of Pertuzumab
Description: The volume of distribution at steady state (Vss), also known as apparent volume of distribution, is a pharmacological, theoretical volume that the total amount of administered drug would have to occupy (if it were uniformly distributed), to provide the same concentration as it currently is in blood plasma.
Time Frame: as for outcome 13
Population: ITT Population; Only participants with non-missing data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 35 | 31
mL | 4452 (26) | 5227 (24)

20. Secondary Outcome: Mean Residence Time (MRT) of Pertuzumab
Description: MRT is the average time that pertuzumab is present in the systemic circulation and is measured in days.
Time Frame: as for outcome 13
Population: ITT Population; Only participants with non-missing data were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Number analyzed (Participants) | 35 | 31
days | 18.1 (42) | 25.7 (77)

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded from the date of Screening until 7 weeks after the last infusion of study treatment.
Arm/Group | Pertuzumab 420 mg - Cohort A | Pertuzumab 1050 mg - Cohort B
Serious Adverse Events (participants affected / at risk) | 9/35 | 6/33
Other Adverse Events (participants affected / at risk) | 28/35 | 24/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab 420 mg - Cohort A (N=35) | Pertuzumab 1050 mg - Cohort B (N=33)
Urinary retention (Renal and urinary disorders) | 3 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Hematolytic Uremic Syndrome (Blood and lymphatic system disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0
Electrocardiogram wave Inversions (Investigations) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Cauda Equina Syndrome (Nervous system disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Hemastemisis (Gastrointestinal disorders) | 0 | 1
Ileus Paralytic (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Central Line Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Metastatic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pertuzumab 420 mg - Cohort A (N=35) | Pertuzumab 1050 mg - Cohort B (N=33)
Diarrhoea (Gastrointestinal disorders) | 18 | 17
Nausea (Gastrointestinal disorders) | 11 | 2
Constipation (Gastrointestinal disorders) | 3 | 1
Flatulence (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 4 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 15 | 4
Asthenia (General disorders) | 3 | 2
Pyrexia (General disorders) | 3 | 1
Influenza Like Illnes (General disorders) | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dysponea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pharyngnolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Backpain (Musculoskeletal and connective tissue disorders) | 5 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 | 4
Arhralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Buttock Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Dysguesia (Nervous system disorders) | 4 | 1
Headache (Nervous system disorders) | 3 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 2
Paraesthesia (Nervous system disorders) | 2 | 1
Rhinitis (Infections and infestations) | 3 | 2
Nasopharyngitis (Infections and infestations) | 3 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 8 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 4
Onychorrhexis (Skin and subcutaneous tissue disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 4 | 0
Dysuria (Renal and urinary disorders) | 2 | 0
Urinary Retention (Renal and urinary disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Ejection Fraction Decreased (Investigations) | 2 | 1

LIMITATIONS AND CAVEATS:
The study was terminated at the time of interim analysis since none of the participants showed a PSA response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.